CLINICAL TRIAL: NCT01683812
Title: Cranial Cup Use for the Correction of Positional Head Shape Deformities in Hospitalized Premature Infants
Brief Title: Cranial Cup Use for Correction of Head Shape Deformities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michele DeGrazia, Director of Nursing Research NICU, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00003465
Record Dates: First submitted 2012-08-29; First posted 2012-09-12 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Dolichocephaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cranial Cup Arm (Experimental): Single arm
  Interventions: Device: Cranial Cup

INTERVENTIONS:
Device: Cranial Cup — Study participants with dolichocephaly will be treated with the Cranial Cup for a minimum 12 hours per day.

SUMMARY:
The purpose of this descriptive study is to provide information on the feasibility of using the cranial cup, a new positioning device, in a small sample of prematurely born infants with elongated head shapes as a result of laying on their abdomens, during the convalescent phase of their hospitalizations.

DETAILED DESCRIPTION:
The cranial cup is a non-invasive, non-restrictive, adjustable orthotic device that grows with the infant and maintains proper body alignment while promoting normal head shape development. While the cranial cup is not yet FDA approved, it is considered a non-significant medical device and it has successfully corrected asymmetric positional head shape deformities in hundreds of healthy newborns less than 4 months of age cared for by the Children's Hospital Boston outpatient plagiocephaly clinic. Additionally preliminary analysis of a prospective randomized controlled trial currently underway suggests that the cranial cup may be useful in prevention of positional head shape deformity in a cohort of hospitalized infants of varying gestational ages. However, the cranial cup has never been used for correction of the most common form of positional head shape deformity in hospitalized premature infants; namely dolichocephaly. Thus, the purpose of this descriptive study is to provide information on the feasibility of using the cranial cup in a small sample of prematurely born infants with dolichocephaly during the convalescent phase of their hospitalizations. Information obtained from this descriptive study will be used to determine if a larger investigation using the cranial cup is warranted in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* Born at < or equal to 35 weeks gestation
* Cleared for participation by healthcare team
* Estimated minimum length of stay >14 days
* Weight >1000 grams (at enrollment)
* Dolichocephalic head shape deformity

Exclusion Criteria:

* Unable to maintain airway patency (anatomical problem)
* Craniofacial anomaly or scalp device, drain or shunt
* Craniosynostosis
* Severe parturitional head shape deformity

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele DeGrazia, PhD, Principal Investigator — Boston Children's Hospital; Aimee Knorr, MD, Principal Investigator — Winchester Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cranial Cup Arm
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cranial Cup Arm
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: weeks] — Corrected Gestational Age at Enrollment
  weeks | 34.6 [30 to 44.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Safety
Description: Nurses will complete daily logs indicating the number of desaturation events (oxygen saturation of < 90 percent for infant corrected to full term or < 87 percent for a premature infant for > 10 seconds) and emesis events (regurgitation of breast milk or formula) during cranial cup device use. The cup's designated use is for at least 12 hours per day. Study duration is at least 14 days and can continue until the infant is discharged. Comparisons will be made for the number of desaturation events and emesis during data analysis.
Time Frame: Logs of cranial cup use and desaturation and emesis events will be recorded for 14 -120 days
Measure: Median (Full Range); unit: count
Arm/Group | Cranial Cup Arm
Number analyzed (Participants) | 23
count
  desaturation events | 7 [0 to 123]
  emesis events | 1 [0 to 8]

2. Secondary Outcome: Cranial Measurement Description
Description: To describe infant head shape, the study will use cranial measurements and laser head scans in a sample of prematurely born Neonatal Intensive Care (NICU) or Special Care Nursery (SCN) patients with dolichocephaly. Cranial measurement used is cranial index, an objective measure that quantifies head shape by dividing the head width (M-L) by length (A-P) then multiplying it by 100%. Measurements and scans will be taken directly following study enrollment and discharge to document head shape pre and post intervention. The discharge measure will be obtained at approximately 2 weeks-4 months of age at hospital discharge.
Time Frame: Using head measurements obtained at timepoint 1 enrollment (baseline, day 1) and at timepoint 2 discharge (14-120 days)
Measure: Median (Full Range); unit: cranial index %
Arm/Group | Cranial Cup Arm
Number analyzed (Participants) | 23
cranial index % | 77.5 [69.8 to 83.9]

ADVERSE EVENTS:
Arm/Group | Cranial Cup Arm
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No